CLINICAL TRIAL: NCT04142853
Title: Walking-related Performance Fatigabitity in People With Multiple Sclerosis: Clinical Profile o
Brief Title: Underlying Causes and Related Factors, and Rehabilitation Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: University of Liege (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: B707201835771
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Persons with MS, dance group (Experimental)
  Interventions: Other: Training intervention + Dance intervention
- Persons with MS, art group (Active Comparator)
  Interventions: Other: Training intervention + Dance intervention

INTERVENTIONS:
Other: Training intervention + Dance intervention — Training intervention + Dance intervention

SUMMARY:
This study will be a cross-sectional observational study, followed by a pilot intervention. The aim of the study is to examine the underlying causes of walking-related performance fatigability, together with other related and influencing factors, to make up a clinical profile of patients with MS showing walking-related performance fatigability. In the second part of the study a pilot intervention will be executed to see if the investigators can improve the clinical status of the MS patients with walking-related performance fatigability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years.
* MS diagnosis according to McDonald Criteria.
* Capable of walking 6 minutes (independent or with unilateral support) without stopping.

Exclusion Criteria:

* Exacerbation or relapse within last 3 months before study
* Other medical condition interfering with walking ability (e.g. cardiac or respiratory diseases, arthritis and fibromyalgia, stroke, Parkinson).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
the Coordination test | Day 1
  Participant is seated with legs strapped in to the mounts and moves legs to the beat of a metronome to assess central motor control.
TST (Triple Stimulation Technique) | day 3
  Technique in which nerves are stimulated to check guidance in the central nervous system
TMS (Transcranial Magnetic Stimulation) | Day 3
  Technique in which nerves are stimulated to check guidance in the central nervous system
the Voluntary Drive test | Day 1
  The participant is seated in a Biodex. While performing a leg extension the Quadriceps muscle is stimulated to check the guidance of electrical signals to the muscles.
the Fatigability Index Legs | Day 1
  Participant is seated in a Biodex and a protocol is performed to establish the muscle strength and muscle endurance of the legs.
Analysis of a Muscle Biopsy | Day 3
  A small piece of muscle tissue of the weakest leg will be biopsied and analyzed in the lab.
the Digit Span | Baseline
  Cognitive test where numbers must be recalled in a certain order to evaluate short term memory
the Digit Span | Week 11
  Cognitive test where numbers must be recalled in a certain order to evaluate short term memory
the Stroop test | Baseline
  Cognitive test to evaluate attention and simultaneous processing of multiple stimuli.
the Stroop test | week 11
  Cognitive test to evaluate attention and simultaneous processing of multiple stimuli.
the Paced Auditory Serial Addition Test (PASAT) | Baseline
  This is a cognitive test where the participant will try to retain certain numbers they hear and do math. Correct answer last 1/3 vs first 1/3
the Paced Auditory Serial Addition Test (PASAT) | Week 11
  This is a cognitive test where the participant will try to retain certain numbers they hear and do math. Correct answer last 1/3 vs first 1/3
the Symbol Digit Modality Test (SDMT) (Cognitive fatigability) | Baseline
  his is a cognitive performance test, substantiated with focus, speed, and visual scanning. Correct answers last 30 seconds vs first 30 seconds
the Symbol Digit Modality Test (SDMT) (Cognitive fatigability) | week 11
  his is a cognitive performance test, substantiated with focus, speed, and visual scanning. Correct answers last 30 seconds vs first 30 seconds
Motor function test (lower limb muscle strength) | Baseline
  This is a motor test to assess the functional lower limb muscle strength. The participant is asked to stand from a seated position and sit down again as fast as possible for five times in a row.
Motor function test (lower limb muscle strength) | week 11
  This is a motor test to assess the functional lower limb muscle strength. The participant is asked to stand from a seated position and sit down again as fast as possible for five times in a row.
25 Foot Walk (T25FW) test | Baseline
  his is a motor test at which the participant is instructed to walk 25 ft (=7,62 meter) as fast and safely as possible. This is a quantitative performance test to assess mobility and leg function.
25 Foot Walk (T25FW) test | week 11
  his is a motor test at which the participant is instructed to walk 25 ft (=7,62 meter) as fast and safely as possible. This is a quantitative performance test to assess mobility and leg function.
Nine Hole Peg Test (NHPT) | Baseline
  This is a motor test to assess the participant's manual skills. This test records the time the participant needs to place 9 pins in the pegboard and remove them again.
Nine Hole Peg Test (NHPT) | week 11
  This is a motor test to assess the participant's manual skills. This test records the time the participant needs to place 9 pins in the pegboard and remove them again.
Fatigability Index Hand | Baseline
  Grip strength will be evaluated through a Jamar dynamometer.
Fatigability Index Hand | week 11
  Grip strength will be evaluated through a Jamar dynamometer.
Activity tracker | Up to 5 days
  A sensor will be placed around the foot and worn by the participant for 5 days and nights to evaluate physical activity and quality of sleep.
Glycocheck | Baseline
  A small camera will be placed under the tongue of the participant and blood vessels will be filmed to determine the quality of the blood vessels and immunity.
Six minute walking test | once during the observational study
  Participant have to walk as far as they can for 6 minutes. Total distance walked and fatigability by comparing first and last minute distance will be calculated.

SECONDARY OUTCOMES:
Fatigue severity scale (FSS) | baseline
  A self-report scale of nine items about fatigue, its severity and how it affects certain activities. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities. It is simple to understand and takes an average of eight minutes to answer
Fatigue severity scale (FSS) | week 11
  A self-report scale of nine items about fatigue, its severity and how it affects certain activities. Answers are scored on a seven point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63. The higher the score, the more severe the fatigue is and the more it affects the person's activities. It is simple to understand and takes an average of eight minutes to answer
Modified Fatigue Impact Scale (MFIS) | baseline
  This is a short questionnaire to evaluate to impact of general fatigue. This questionnaire measures the effects of fatigue on three levels: physical, cognitive and psychosocial. The MFIS is a 21-item questionaire, scale 0 (never)-4 (always), scale range 0-40
Modified Fatigue Impact Scale (MFIS) | week 11
  This is a short questionnaire to evaluate to impact of general fatigue. This questionnaire measures the effects of fatigue on three levels: physical, cognitive and psychosocial.The MFIS is a 21-item questionaire, scale 0 (never)-4 (always), scale range 0-40
Fatigue Scale of Motor and Cognitive Functions (FSMC) | baseline
  This is a short questionnaire to cognitive and motor fatigue in people with MS. The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue). Two subscales (mental and physical fatigue) can be made. Items included in the subscale mental are 1-4-7-8-11-13-15-17-18-20 and items included in the subscale physical are 2-3-5-6-9-10-12-14-16-19.
Fatigue Scale of Motor and Cognitive Functions (FSMC) | week 11
  This is a short questionnaire to cognitive and motor fatigue in people with MS. The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue). Two subscales (mental and physical fatigue) can be made. Items included in the subscale mental are 1-4-7-8-11-13-15-17-18-20 and items included in the subscale physical are 2-3-5-6-9-10-12-14-16-19.
Hospital Anxiety and Depression Scale (HADS) | baseline
  This is a short questionnaire that evaluates symptoms of anxiety and depression in daily life. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression..
Hospital Anxiety and Depression Scale (HADS) | Week 11
  This is a short questionnaire that evaluates symptoms of anxiety and depression in daily life. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
The Sleep Condition Indicator (SCI) | baseline
  This is a short questionnaire to evaluate sleeping pattern and potential sleeping disorders. The Sleep Condition Indicator (SCI) is an eight-item rating scale (4-0) that was developed to screen for insomnia disorder based on DSM-5 criteria.
The Sleep Condition Indicator (SCI) | week 11
  This is a short questionnaire to evaluate sleeping pattern and potential sleeping disorders. The Sleep Condition Indicator (SCI) is an eight-item rating scale (4-0) that was developed to screen for insomnia disorder based on DSM-5 criteria.
Social Role Participation Questionnaire (SRPQ) | baseline
  This is a short questionnaire to evaluate social participation. scale 1 (not important) - 5(very important)
Social Role Participation Questionnaire (SRPQ) | week 11
  This is a short questionnaire to evaluate social participation. scale 1 (not important) - 5 (very important)
pre-interventionMSWS-12 score | baseline
  short questionnaire to map out walking difficulties in daily living. The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
  A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100. Walking improvement on the MSWS-12 is indicated by negative change scores.
post-interventionMSWS-12 score | baseline
  short questionnaire to map out walking difficulties in daily living. The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
  A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100. Walking improvement on the MSWS-12 is indicated by negative change scores.
pre-interventionMSWS-12 score | week 11
  short questionnaire to map out walking difficulties in daily living. The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
  A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100. Walking improvement on the MSWS-12 is indicated by negative change scores.
post-interventionMSWS-12 score | week 11
  short questionnaire to map out walking difficulties in daily living. The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
  A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100. Walking improvement on the MSWS-12 is indicated by negative change scores.
Multiple Sclerosis Impact Scale (MSIS-29) | Baseline
  This is a short self-report questionnaire used to assess the day-to-day life in the past two weeks. This questionnaire has a physical and psychological scale. The MSIS-29 is a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease on daily function (worse health).
  The physical impact score is computed by summing items number 1-20 inclusive. This score can then be transformed to a score on a scale of 0 -100
Multiple Sclerosis Impact Scale (MSIS-29) | week 11
  This is a short self-report questionnaire used to assess the day-to-day life in the past two weeks. This questionnaire has a physical and psychological scale. The MSIS-29 is a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5"extremely". Each of the two scales are scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates greater impact of disease on daily function (worse health).
  The physical impact score is computed by summing items number 1-20 inclusive. This score can then be transformed to a score on a scale of 0 -100
Short Form Health survey (SF-36) | Baseline
  questionnaire to measure health status. The Optum® SF-36v2® Health Survey asks 36 questions to measure functional health and well-being from the patient's point of view. It is a practical, reliable and valid measure of physical and mental health that can be completed in five to ten minutes.
Short Form Health survey (SF-36) | week 11
  questionnaire to measure health status. The Optum® SF-36v2® Health Survey asks 36 questions to measure functional health and well-being from the patient's point of view. It is a practical, reliable and valid measure of physical and mental health that can be completed in five to ten minutes.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Hasselt University, Hasselt
  - Centre Hospitalier Universitaire de Liège, Liège

REFERENCES:
- [Derived] Goetschalckx M, Van Geel F, Meesen R, Triccas LT, Geraerts M, Moumdjian L, Feys P. Interlimb Coordination Performance in Seated Position in Persons With Multiple Sclerosis: Reduced Amplitude Over 6 min and Higher Coordination Variability in Persons With Walking Fatigability. Front Hum Neurosci. 2021 Oct 20;15:765254. doi: 10.3389/fnhum.2021.765254. eCollection 2021. PMID 34744669